CLINICAL TRIAL: NCT00416741
Title: Assessing The Treatment Effect in Metabolic Syndrome Without Perceptible diabeTes (ATTEMPT)
Acronym: ATTEMPT
Status: Completed | Type: Observational
Sponsor: Hellenic Atherosclerosis Society (Other)
Responsible Party: V.G. Athyros, MD Study Administrator, HellenicAS
Other Study IDs: HAS-01-231206
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Obesity; Hyperlipidemia; High blood pressure; Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hyperlipidemias; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 Usual Care-Lifestyle counseling: Metabolic syndrome
  Interventions: Behavioral: Implementation of guidelines
- 2 Intensive care-Lifestyle counseling: Metabolic Syndrome Implementation of guidelines
  Interventions: Behavioral: Implementation of guidelines

INTERVENTIONS:
Behavioral: Implementation of guidelines — Attaining targets for LDL cholesterol, arterial blood pressure, fasting [plasma flucose

SUMMARY:
The objective of this protocol is to improve awareness, treatment, and control of metabolic syndrome, within primary prevention of cardiovascular disease, by implementing guidelines, after training of the participating physicians.

DETAILED DESCRIPTION:
Physicians from 20 hospitals or health centres (primary and secondary health care settings) were trained to implement guidelines in treating metabolic syndrome.

There will be a baseline recording of patients with metabolic syndrome and then physicians will have to complete a one page form (by ticking pre-specified boxes) about the baseline status of the patients and will have to report the measures they took to improve awareness, treatment, and effective control of the metabolic syndrome. With 6 month intervals (up to 36 months at study completion) physicians will have to complete the same form. Previous training of physicians and the fact that they will have to report their success in treating metabolic syndrome will hopefully contribute to an increase in number of patients with the syndrome at treatment targets, and will minimise the target organ damage (i.e cardiovascular disease). The estimated 10-year reduction in coronary heart disease risk will be evaluated by a comparison of this risk (as evaluated by a risk engine, i.e. PROCAM) at the 6th month and at study completion with that of baseline.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome (NCEP ATP III Definition modified to AHA/NHLBI definition)

Exclusion Criteria:

* Pregnancy
* Lactation
* Malignancies with small life expectancy
* Unwillingness to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metabolic Syndrome (NCEP ATP III Definition modified to AHA/NHLBI definition)
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2005-02; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios G Athyros, MD, Study Chair — Clinical Trials Chair of Hellenic Atherosclerosis Society; Moses - Elisaf, MD, Study Director — Clinical Trials Director of Hellenic Atherosclerosis Society
Locations (1):
- Hellenic Atherosclerosis Society, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Background] Athyros VG, Ganotakis ES, Elisaf MS, Liberopoulos EN, Goudevenos IA, Karagiannis A; GREECE-METS Collaborative Group. Prevalence of vascular disease in metabolic syndrome using three proposed definitions. Int J Cardiol. 2007 Apr 25;117(2):204-10. doi: 10.1016/j.ijcard.2006.04.078. Epub 2006 Jul 18. PMID 16854482
- [Background] Daskalopoulou SS, Athyros VG, Kolovou GD, Anagnostopoulou KK, Mikhailidis DP. Definitions of metabolic syndrome: Where are we now? Curr Vasc Pharmacol. 2006 Jul;4(3):185-97. doi: 10.2174/157016106777698450. PMID 16842136
- [Background] Athyros VG, Ganotakis ES, Bathianaki M, Monedas I, Goudevenos IA, Papageorgiou AA, Papathanasiou A, Kakafika AI, Mikhailidis DP, Elisaf M; MetS-Greece Collaborative Group. Awareness, treatment and control of the metabolic syndrome and its components: a multicentre Greek study. Hellenic J Cardiol. 2005 Nov-Dec;46(6):380-6. PMID 16422124
- [Background] Athyros VG, Mikhailidis DP, Papageorgiou AA, Didangelos TP, Peletidou A, Kleta D, Karagiannis A, Kakafika AI, Tziomalos K, Elisaf M. Targeting vascular risk in patients with metabolic syndrome but without diabetes. Metabolism. 2005 Aug;54(8):1065-74. doi: 10.1016/j.metabol.2005.03.010. PMID 16092057
- [Derived] Athyros VG, Karagiannis A, Ganotakis ES, Paletas K, Nicolaou V, Bacharoudis G, Tziomalos K, Alexandrides T, Liberopoulos EN, Mikhailidis DP; Assessing The Treatment Effect in Metabolic syndrome without Perceptible diabeTes (ATTEMPT) Collaborative Group. Association between the changes in renal function and serum uric acid levels during multifactorial intervention and clinical outcome in patients with metabolic syndrome. A post hoc analysis of the ATTEMPT study. Curr Med Res Opin. 2011 Aug;27(8):1659-68. doi: 10.1185/03007995.2011.595782. Epub 2011 Jun 30. PMID 21714711
- [Derived] Athyros VG, Ganotakis E, Kolovou GD, Nicolaou V, Achimastos A, Bilianou E, Alexandrides T, Karagiannis A, Paletas K, Liberopoulos EN, Tziomalos K, Petridis D, Kakafika A, Elisaf MS, Mikhailidis DP; Assessing The Treatment Effect in Metabolic Syndrome Without Perceptible Diabetes (ATTEMPT) Collaborative. Assessing the treatment effect in metabolic syndrome without perceptible diabetes (ATTEMPT): a prospective-randomized study in middle aged men and women. Curr Vasc Pharmacol. 2011 Nov;9(6):647-57. doi: 10.2174/157016111797484080. PMID 21476961
- [Derived] Chimonas T, Athyros VG, Ganotakis E, Nicolaou V, Panagiotakos DB, Mikhailidis DP, Elisaf M; Assessing the Treatment Effect in Metabolic Syndrome Without Perceptible diabeTes (ATTEMPT) Collaborative Group. Cardiovascular risk factors and estimated 10-year risk of fatal cardiovascular events using various equations in Greeks with metabolic syndrome. Angiology. 2010 Feb-Mar;61(1):49-57. doi: 10.1177/0003319709351873. PMID 20034959
- See also: PMID: 21476961-Assessing The Treatment Effect in Metabolic Syndrome without Perceptible Diabetes (ATTEMPT): A Prospective-Randomized Study in Middle Aged Men and Women. — http://www.ncbi.nlm.nih.gov/pubmed?term=athyros